CLINICAL TRIAL: NCT05704907
Title: Diagnostic Performance of Dual Energy CT for the Detection of Gallbladder Gallstones
Acronym: DUAL-GB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/743
Record Dates: First submitted 2023-01-17; First posted 2023-01-30 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Gallstone
Keywords: abdominal and pelvic scan; abdominal Ultrasound
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gallblader ultrasound (Other)
  Interventions: Other: gallbladder ultrasound

INTERVENTIONS:
Other: gallbladder ultrasound — gallbladder ultrasound

SUMMARY:
To assess diagnostic performance of Dual Energy CT fo gallblader gallstone detection.

DETAILED DESCRIPTION:
Detection of gallbladder gallstone using Dual Energy CT compare to gallblader ultrasound (gold standard).

All patients who undergo dual-energy CT scans will undergo abdominal ultrasound for gallstones.

Performance of CT to conventionnal KeV will be compare to low Kev monoenergetic reconstruction, and Effective Z.

Expected duration of inclusion 3-6 months. No follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patient referred to the radiology department for an abdominal CT for abdominal pain, suspicion of cholangitis, cholecystitis, migration of stones, acute pancreatitis, suspicion of perforated ulcer in the emergency setting.
* Non-objection of the subject to participate in the study
* Affiliation to a French social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Cholecystectomy
* Legal incapacity or limited legal capacity, legal safeguard
* Pregnant women
* Subject unlikely to cooperate in the study and/or low cooperation anticipated by the investigator
* Subject being in the exclusion period of another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Gallstone detection using Dual Energy CT | Day 0
  Number - size of gallstones

SECONDARY OUTCOMES:
Gallstone detection using reconstruction to conventionnal KeV. | Day 0
  Number - size of gallstones

CONTACTS AND LOCATIONS:
Overall Officials: Paul CALAME, MD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided